CLINICAL TRIAL: NCT00692757
Title: Comparative Study of Two Antiseptics Solutions for the Prevention of Surgical Site Infection
Brief Title: Wound Antiseptic Study With Hypochlorous Acid & Iodopovidone
Acronym: WASH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Tecnológica de Pereira (Other)
Collaborators: Hospital Universitario San Jorge de Pereira (HUSJ) (Unknown)
Responsible Party: Juliana Buitrago Jaramillo, Universidad Tecnológica de Pereira
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5-07-9
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Surgical Site Infection
Keywords: Hypochlorous Acid; Colony forming units; surgical site infection; nosocomial infection; bacterial bioburden; wound healing
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection | interventions — Hypochlorous Acid; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Hypochlorous acid
  Interventions: Drug: Hypochlorous acid
- B (Active Comparator): Iodopovidone
  Interventions: Drug: Iodopovidone

INTERVENTIONS:
Drug: Hypochlorous acid — Hypochlorous acid for preoperative scrubbing to prevent surgical site infection in spray
  Other Names: NVC-101 NovaBay Pharmaceuticals, Inc, Emeryville, CA
  Arms: A
Drug: Iodopovidone — Iodopovidone
  Arms: B

SUMMARY:
The purpose of this study is to determine whether hypochlorous acid is an effective antiseptic agent to prevent surgical site infection.

DETAILED DESCRIPTION:
A topical antimicrobial that decrease the bacterial bioburden of surgical wounds without impairing the wound's ability to heal is a need. A stabilized form of hypochlorous acid has been demonstrated in vitro and in animal studies to possess properties that could fulfill these criteria but it is imperative to assess its efficacy and safety in humans.

To assess hypochlorous acid efficacy and safety, it was designed a clinical controlled randomized trial to compare hypochlorous acid to iodopovidone, the gold standard, in preoperative scrub of surgical area.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old, who are going to be operated
* Classification of surgical wounds according to the National Research Council as class I or II
* Risk index classification of the American Society of Anaesthesiology (ASA) as ASA 1 or 2

Exclusion Criteria:

* Patients requiring mesh or prosthesis or orthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-01 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection rates | until one month (weekly)

SECONDARY OUTCOMES:
Decreasing Colony Forming Unit count (CFU/mL) after using the skin topic antiseptic in surgical site | one week

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Buitrago, MD.,MSc, Principal Investigator — Universidad Tecnológica de Pereira
Locations (1):
- Hospital Universitario San Jorge (HUSJ), Pereira, Risaralda Department, Colombia

REFERENCES:
- [Background] Selkon JB, Cherry GW, Wilson JM, Hughes MA. Evaluation of hypochlorous acid washes in the treatment of chronic venous leg ulcers. J Wound Care. 2006 Jan;15(1):33-7. doi: 10.12968/jowc.2006.15.1.26861. PMID 16669304
- [Background] Robson MC, Payne WG, Ko F, Mentis M, Donati G, Shafii SM, Culverhouse S, Wang L, Khosrovi B, Najafi R, Cooper DM, Bassiri M. Hypochlorous Acid as a Potential Wound Care Agent: Part II. Stabilized Hypochlorous Acid: Its Role in Decreasing Tissue Bacterial Bioburden and Overcoming the Inhibition of Infection on Wound Healing. J Burns Wounds. 2007 Apr 11;6:e6. PMID 17492051
- [Background] Wang L, Bassiri M, Najafi R, Najafi K, Yang J, Khosrovi B, Hwong W, Barati E, Belisle B, Celeri C, Robson MC. Hypochlorous acid as a potential wound care agent: part I. Stabilized hypochlorous acid: a component of the inorganic armamentarium of innate immunity. J Burns Wounds. 2007 Apr 11;6:e5. PMID 17492050